CLINICAL TRIAL: NCT03522025
Title: A Prospective, Multicenter, Randomised Study to Evaluate the Fixation of Cemented and Cementless Design of GMK-UNI Anatomical Knee Prosthesis.
Brief Title: GMK-UNI Anatomical UKA: Fixation of Cemented vs Cementless Designs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-01677
Record Dates: First submitted 2018-04-27; First posted 2018-05-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GMK-UNI cemented fixation prosthesis (Active Comparator): Unicompartmental Knee Arthroplasty (UKA)
  Interventions: Device: Unicompartmental Knee Arthroplasty (UKA)
- GMK-UNI cementless fixation prosthesis (Experimental): Unicompartmental Knee Arthroplasty (UKA)
  Interventions: Device: Unicompartmental Knee Arthroplasty (UKA)

INTERVENTIONS:
Device: Unicompartmental Knee Arthroplasty (UKA) — Unicompartmental Knee Arthroplasty (UKA) is a less invasive treatment option compared to Total Knee Arthroplasty (TKA) for patients with primary anteromedial knee osteoarthritis.

SUMMARY:
Unicompartmental knee arthroplasty (UKA) is the principal surgical alternative to the total knee arthroplasty (TKA) in patients with end-stage unicompartmental tibiofemoral osteoarthritis (OA) of the knee. The current comparative randomized study aims to evaluate the fixation of cemented and cementless designs of GMK-UNI unicompartmental knee prosthesis over a 5-year time period.

DETAILED DESCRIPTION:
The Primary objective is to compare the quality of fixation of cemented and cementless designs of GMK-UNI unicompartmental knee replacement at 2 years of follow-up.

The Secondary objectives include the evaluation of the patient improvement (subjective and objective) using the new Knee Society Score (KSS); the patient's anterior pain following UKA and any eventual patella-femoral disorder; Implant survival rate using the Kaplan Meier analysis; Post-op radiological findings and Adverse Events.

The Primary outcome aims to compare the occurrence of radiolucency's lines (both partial and complete) between the two study groups. Secondary outcomes include New KSS, OKS, Kaplan Meier analysis and stability and fixation of UNI prosthesis.

All patients who meet the inclusion criteria to take part in the current clinical study will be invited to participate before the surgery.

Subjects will be randomized during the screening; half of them will receive the cemented GMK-UNI anatomical UKA and the other half the cementless GMK-UNI anatomical UKA.

Clinical data will be recorded on CRF at those time-points:

* Before the surgery
* During the surgery
* After the surgery at 3 months, 1, 2, 3 and 5 years.

ELIGIBILITY:
Inclusion criteria:

* Patients with end-stage unicompartmental tibiofemoral osteoarthritis (OA) of the knee that meet the indications for use according to Medacta implants included in this study (on-label use);
* Those suffering from unilateral osteoarthritis or osteonecrosis of the medial compartment;
* Frontal deformity < 10° (evaluated on weight-bearing long-axis x-rays);
* Flexion contracture < 10°;
* Intact ligaments;
* Patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to the patient's surgery;
* Patient's age over 18 years old;
* Patient with BMI < 40 kg/m2;
* Patients must be willing to comply with the pre and post-operative evaluation schedule.

Exclusion criteria:

* Patients with one or more medical conditions identified as a contraindication defined by the labelling on any Medacta implants used in this study;
* Any patient who cannot or will not provide informed consent for participation in the study;
* Patients who need to undergo lateral unicompartmental knee arthroplasty;
* Patients who need a revision surgery;
* Patients who need a patella-femoral joint prosthesis;
* Patients who had previously undergone high tibial osteotomy or ACL reconstruction;
* Patients with BMI ≥ 40 kg/m2;
* Patients unable to understand and take action;
* Any case not described in the inclusion criteria;
* Patients aged under 18 years;

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the occurrence of radiolucency's lines | 5 yrs
  Compare occurrence of radiolucency's lines (both partial and complete)between the two study groups

SECONDARY OUTCOMES:
Anterior Knee Pian Scale (Kujala score) | pre-op; 3months;1,2,3,5 yrs
  It's a 13-item knee specific self-report questionnaire. It documents response to 6 activities associated with anterior knee pain as well as symptoms such as limp, inability to weight bear through the affected limp, swelling...). It asks about duration of symptoms and limbs affected. Max score is 100 and lower scores indicate greater pain/disability. Scoring is hierarchical using various types of categorisation including "no difficulty-unable " and "no pain-severe pain". It is easy to understand and takes few minutes to complete.It has a good test-retest reliability.
Implant survival rate using Kaplan Meier analysis | 5 yrs
  Implant survival rate
Recording of adverse events | Throughout the study
  Any complication occurred during the study
Oxford Knee Score | Pre-op;3month;1,2,3,5yrs
  The Oxford Knee Score (OKS) is a 12-item patient-reported PRO specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty).Each question is scored from 1 to 5, with 1 representing best outcome/least symptoms. Scores from each question are added so the overall score is from 12 to 60 (12 being the best outcome). The overall score for the OKS is acquired by simply summing the scores received for individual questions.
New Knee Society Score | Pre-op:3months;1,2,3,5 yrs
  The new KSS System is a validated and responsive method for assessing objective and subjective outcomes after total and partial knee arthroplasty.It includes versions to be admninstered pre-op and post-op.It has an initial assessment of demographic deatils. The objective knee score includes VAS score of pain walking on level ground and on stairs or inclines, as well as ROM, an assessment of alignment, ligament stability along with deductions for flexion contracture or extensor lag. Pts then record their satisfaction, functional activities and expectations. It consists of 4 subscales: 1) objective knee score (7 items;100 points); 2) Satisfaction Score (5 items; 40 points);3) Expectation Score (3 items; 15 points); 4) Functional Activity Score (19 items; 100 points)
Stability and fixation of unicompartmental prosthesis | 5 yrs
  To evaluate the stability and fixation of the prosthesis

CONTACTS AND LOCATIONS:
Locations (5):
- France (4):
  - Clinique Saint Vincent de Paul, Bourgoin, France
  - Clinique du Mail, La Rochelle, France
  - Centre Orthéo, Espace Fauriel, Saint-Etienne, France
  - CHP Saint-Grégoire, Saint-Grégoire, France
- Dr. Näder Helmy, Solothurn, Switzerland, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided